CLINICAL TRIAL: NCT03446638
Title: iCare 2: Personalized Genomic Mutation Informed Treatment of Patients With Myelodysplastic Syndromes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: administratively withdrawn
Sponsor: University of Florida (Other)
Collaborators: Gateway for Cancer Research (Other); Cellworks Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iCare 2; OCR17918 (Other: UF OnCore); IRB201702867 (Other: University of Florida)
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: myelodysplastic syndromes; MDS; computational biology; relapsed; refractory
MeSH Terms: conditions — Myelodysplastic Syndromes; Recurrence | interventions — Cytarabine; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Computational Biology-Informed Treatment (Experimental): Patients randomized to this arm will receive an FDA-approved drug or combination of drugs predicted to have a therapeutic effect based on their individual MDS disease genetic profile by a computational biology simulation software program. The specific drug or combination of drugs that a patient on this arm will receive will be decided jointly by a molecular oncology board comprised of physicians, pharmacists, and nurse coordinators and the treating physician. Patients will receive a minimum of 2 months and a maximum of 4 months of treatment with the selected drug or combination of drugs.
  Interventions: Drug: FDA-approved drug or combination of drugs; Device: Computational biology simulations software
- Standard of Care Treatment (Active Comparator): Patients randomized to this arm will receive either one of three standard of care treatment regimens of the treating physician's choice (low-dose cytarabine, 7 + 3 induction, or FLAG induction) or supportive care alone. Patients will receive a minimum of 2 months and a maximum of 4 months of the selected treatment regimen or of supportive care alone.
  Interventions: Drug: FLAG induction; Drug: 7 + 3 induction; Drug: Low-dose cytarabine; Other: Supportive care alone

INTERVENTIONS:
Drug: FDA-approved drug or combination of drugs — Patients assigned to this arm will receive an FDA-approved drug or combination of drugs. Dosing and treatment schedule will follow the package insert for the selected drug(s).
  Arms: Computational Biology-Informed Treatment
Drug: FLAG induction — Patients will receive 30 mg/m2 per day intravenously of fludarabine for 5 days and 2000 mg/m2 per day intravenously of cytarabine for 5 days. 5 mg/kg per day of granulocyte colony stimulating factor (G-CSF) may be given subcutaneously beginning on Day 1 of each treatment until absolute granulocyte count > 500/ microliter for 3 days.
  Arms: Standard of Care Treatment
Drug: 7 + 3 induction — Patients will receive 100-200 mg/m2 per day intravenously of cytarabine for 7 days, plus either 45-60 mg/m2 per day intravenously of daunorubicin or 9-12 mg/m2 per day intravenously of idarubicin for 3 days.
  Arms: Standard of Care Treatment
Drug: Low-dose cytarabine — Patients will receive 20 mg/m2 per day subcutaneously of cytarabine for 10 days every 28 days.
  Arms: Standard of Care Treatment
Other: Supportive care alone — Patients will receive one or more of the following: blood product transfusions, antibiotics, granulocyte colony-stimulating factor (G-CSF), erythropoietic stimulating factors, and iron chelation.
  Arms: Standard of Care Treatment
Device: Computational biology simulations software — Genetic testing results for each patient randomized to this arm will be used by a computational biology simulations software program to generate a personalized map of dysregulated metabolic pathways contributing to the patient's disease. This map will then be used to digitally screen for potentially therapeutic FDA-approved drugs or drug combinations to target the dysregulated metabolic pathways.
  Arms: Computational Biology-Informed Treatment

SUMMARY:
This open-label, randomized, parallel group phase II study will investigate the efficacy of computational biology-informed treatment vs. standard of care treatment for patients with relapsed or refractory myelodysplastic syndromes (MDS).

DETAILED DESCRIPTION:
It is hypothesized that personalized treatment informed by computational biology simulation technology will improve treatment outcomes for patients with relapsed or refractory MDS.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Must be at least 18 years of age
* Diagnosis of MDS, as defined by World Health Organization (WHO) 2008, that has relapsed after any duration of time from last best response or is refractory to induction therapy (defined as 4 cycles of treatment with a hypomethylating agent, 2 cycles of lenalidomide, 1 cycle of low intensity chemotherapy, or 1 cycle of high intensity chemotherapy)
* ECOG performance status of 0-2
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) may participate, provided they meet the following conditions:

  1. Must agree to use physician-approved contraceptive methods (e.g., abstinence, intrauterine device, oral contraceptive, double barrier device) throughout the study and for 3 months following the last dose of study treatment; and
  2. Must have a negative serum or urine pregnancy test within 7 days prior to beginning treatment on this trial
* Males with female partners of child-bearing potential must agree to use physician approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 6 months following the last dose of study treatment.

Exclusion Criteria:

* Must not have acute myeloid leukemia (AML), as defined by WHO 2008
* Pregnant and nursing subjects are excluded because the effects of study treatments on a fetus or nursing child are unknown
* Must not have had treatment with any anti-cancer therapy (investigational or standard) within the previous 21 days prior to the first dose of study drug or less than full recovery (no worse than CTCAE v4.0 grade 1) from the clinically significant toxic effects of that treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Difference in overall response, as measured by International Working Group (IWG) 2006 criteria for response in MDS | 4 months
  Difference in overall response (number of patients who achieve complete response, partial response, stable disease, or hematologic improvement per IWG 2006 criteria) between patients treated with computational biology-informed therapy vs. those treated with standard of care regimens

SECONDARY OUTCOMES:
Difference in safety and feasibility, as measured by CTCAE v4.0 criteria | 5 months
  Difference in safety and feasibility, as measured by CTCAE v4.0 criteria, between patients treated with computational biology-informed treatment and those who receive a standard of care regimen
Difference in time to death between patients treated with computational biology-informed therapy and those treated with standard of care regimens | 3 years
Difference in time to progression to acute myeloid leukemia (AML), as measured by IWG 2006 criteria for response in MDS, between patients treated with computational biology-informed therapy and those treated with standard of care regimens | 4 months
Difference in time to disease relapse, as measured by IWG 2006 criteria for response in MDS, between patients treated with computational biology-informed therapy and those treated with standard of care regimens | 4 months
Difference in time to best response, as measured by IWG 2006 criteria for response in MDS, between patients treated with computational biology-informed therapy and those treated with standard of care regimens | 4 months
Difference in change in myeloblast percentage between patients treated with computational biology-informed therapy and those treated with standard of care regimens | 4 months
Difference in blood transfusion rate between patients treated with computational biology-informed therapy and those treated with standard of care regimens | 7 months

OTHER OUTCOMES:
Differences in mutant allele frequencies between patients treated with computational biology-informed therapy and those treated with standard of care regimens | 4 months
Laboratory correlations between computational model and actual intracellular pathway activation status | 4 months
Clinical correlations between pharmacogenotypes and drug efficacy (as measured by IWG 2006 criteria for response in MDS) | 4 months
Clinical correlations between pharmacogenotypes and drug-related adverse events (as measured by CTCAE v4.0 criteria) | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cogle, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States